CLINICAL TRIAL: NCT05548530
Title: Analysis of Related Factors of Hematoma Morphology in Patients With Cerebral Hemorrhage and Prognosis Analysis of Different Regimens for Cerebral Hemorrhage
Brief Title: Prognostic Analysis of Different Treatment Options for Cerebral Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Zhaoxu，MD, Principal Investigator, The Affiliated Hospital Of Guizhou Medical University
Other Study IDs: JZSJK0828
Record Dates: First submitted 2022-08-31; First posted 2022-09-21 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Brain Hemorrhage
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Decompressive Craniectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stereotactic intracranial hematoma puncture treatment group: Check the CT slice of the patient's brain, find out the patient's largest hematoma level, measure the coordinates of the puncture center, locate and mark the skull surface according to the measured coordinates, select the puncture point under the stereotaxic instrument, Mainly avoid important blood vessels, nerves and functional areas. Use an electric drill to drill the puncture needle into the center of the hematoma, and slowly aspirate the hematoma from the side hole until the suction stops when there is resistance. The residual hematoma in CT and the location of the drainage tube were determined, and the position of the puncture needle was adjusted for the situation of brain CT. After the operation, according to the re-examination of cranial CT, urokinase was injected into the hematoma cavity through the drainage tube to dissolve the residual hematoma, and the operation process strictly followed aseptic operation.
  Interventions: Procedure: Stereotactic intracranial hematoma puncture
- drug treatment group: General treatment: Based on high-level nursing care and close and continuous attention to the patient's vital signs, the patient is instructed to stay in bed continuously, give oxygen, and instruct the patient to avoid emotional agitation, etc. ②Special treatment: use hemostatic drugs, control blood pressure to prevent rebleeding, control blood sugar, control body temperature, anti-epilepsy, prevent infection, dehydration and lower intracranial pressure, etc. Multisystem complications such as tract hemorrhage should be actively managed.
- decompressive craniectomy treatment group: Prior to the procedure, all patients obtained endotracheal intubation under general anesthesia following the informed consent provided by their family members. Upon identifying the hematoma's location through CT imaging, the surgeon made a linear or horseshoe-shaped incision on the scalp and subsequently opened the dura mater after creating a bone flap. The hematoma was punctured using a brain needle, allowing for effective decompression. The cerebral cortex was incised along the cerebral gyri, facilitating the separation of brain tissue to eliminate residual hematoma. Once hemostasis was ensured within the operative area, a silicone drainage tube was inserted, and the cranial bone flap was restored to its original position. In cases of severe brain edema or cerebral herniation, bone flap decompression was performed.
  Interventions: Procedure: decompressive craniectomy
- Neuroendoscopic treatment group: The patient's preoperative CT and MR imaging data were fused with a neuronavigation system to avoid important functional areas and select the closest point of the hematoma to the cortex as the location point. Routine craniotomy was performed with a 2*3 cm bone window, the puncture direction was repositioned by neuronavigation, the sheath was placed at the center of the hematoma, the core was removed, the endoscope was gradually aspirated, and the bleeding was stopped with electrocoagulation if there was considerable active bleeding. A drainage tube was placed, the bone flap was reset after surgery, and the scalp was sutured.
  Interventions: Procedure: Neuroendoscopic

INTERVENTIONS:
Procedure: Stereotactic intracranial hematoma puncture — Check the CT scan of the patient's brain, find out the largest hematoma level of the patient, measure the coordinates of the puncture center, locate and mark the skull surface according to the coordinates obtained from the measurement, select the puncture point under the stereotaxic instrument, and mainly avoid important blood vessels , nerves and functional areas. Use an electric drill to drill the puncture needle into the center of the hematoma, and slowly aspirate the hematoma from the side hole until the suction stops when there is resistance. The residual hematoma in CT and the location of the drainage tube were determined, and the position of the puncture needle was adjusted for the situation of brain CT. After the operation, according to the re-examination of cranial CT, urokinase was injected into the hematoma cavity through the drainage tube to dissolve the residual hematoma, and the operation process strictly followed aseptic operation.
  Groups: Stereotactic intracranial hematoma puncture treatment group
Procedure: decompressive craniectomy — Prior to the procedure, all patients obtained endotracheal intubation under general anesthesia following the informed consent provided by their family members. Upon identifying the hematoma's location through CT imaging, the surgeon made a linear or horseshoe-shaped incision on the scalp and subsequently opened the dura mater after creating a bone flap. The hematoma was punctured using a brain needle, allowing for effective decompression. The cerebral cortex was incised along the cerebral gyri, facilitating the separation of brain tissue to eliminate residual hematoma. Once hemostasis was ensured within the operative area, a silicone drainage tube was inserted, and the cranial bone flap was restored to its original position. In cases of severe brain edema or cerebral herniation, bone flap decompression was performed.
  Groups: decompressive craniectomy treatment group
Procedure: Neuroendoscopic — The patient's preoperative CT and MR imaging data were fused with a neuronavigation system to avoid important functional areas and select the closest point of the hematoma to the cortex as the location point. Routine craniotomy was performed with a 2*3 cm bone window, the puncture direction was repositioned by neuronavigation, the sheath was placed at the center of the hematoma, the core was removed, the endoscope was gradually aspirated, and the bleeding was stopped with electrocoagulation if there was considerable active bleeding. A drainage tube was placed, the bone flap was reset after surgery, and the scalp was sutured.
  Groups: Neuroendoscopic treatment group

SUMMARY:
To analyze the influence of early hematoma morphology on hematoma expansion, optimize the treatment plan for cerebral hemorrhage, and guide the treatment of patients with cerebral hemorrhage in combination with clinical practice.

DETAILED DESCRIPTION:
Intracerebral hemorrhage refers to the hemorrhage caused by the rupture of blood vessels in the non-traumatic brain parenchyma, accounting for 20% to 30% of all strokes, with an acute mortality rate of 30% to 40%. Different degrees of movement disorders, language disorders, etc. will be left behind. It is of great clinical significance to deeply explore the relevant factors and effective treatment plans for the evolution of cerebral hemorrhage. 30% of hematomas can still have active bleeding within 20 hours of onset. The INTERACT test defines hematoma expansion as 24-48 hours of repeated non-enhanced CT. The increase in hematoma volume >12.5ml or 33% of the original volume is the cause of neurological deterioration and abnormality. An important cause of poor prognosis, studies have confirmed that irregular hematoma morphology is a strong predictor of hematoma expansion. Treatment of cerebral hemorrhage currently includes medical treatment and surgical treatment. Surgical treatment has become an important method for the treatment of ICH due to its advantages of rapid removal of hematoma, relief of high intracranial pressure, and release of mechanical compression. However, whether surgery can reduce the mortality of patients with cerebral hemorrhage and improve neurological damage is still controversial. Surgical operations include dstereotactic intracranial hematoma puncture and drainage, decompressive craniectomy , neuroendoscopic. Currently, there are large randomized controlled trials at home and abroad on minimally invasive hematoma evacuation. The treatment of spontaneous intracerebral hemorrhage is safe, but the effectiveness of minimally invasive surgery is unclear due to inconsistent bleeding volume, surgical trauma, and hematoma morphology.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Intracerebral hemorrhage was diagnosed by head CT examination;

Exclusion Criteria:

1. Multiple intracranial hemorrhage;
2. Intracranial hemorrhage caused by intracranial tumor, aneurysm, trauma, infarction or other lesions;
3. Coagulation disorders or a history of taking anticoagulants;
4. Infectious meningitis, systemic infection;
5. History of severe stroke, heart, kidney, liver and lung dysfunction in the past;
6. Severe brain herniation (mydriasis, respiratory and circulatory failure);
7. Incomplete or missing basic data or follow-up information in the hospital.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inpatients admitted to the Emergency Neurology Department of the Affiliated Hospital of Guizhou Medical University from January 1, 2014 to August 31, 2022 were collected. According to the head CT at the time of admission, they were divided into the hematoma rule group and the hematoma irregular group
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematoma expansion rate 24 hours after onset | 24 hours of onset
  The number of cases with enlarged hematoma after re-examination of head CT after 24 hours
90-day Modified Rankin Rating Scale score; | 90-day
  Modified Rankin Rating Scale score at 90 days after discharge，0-3 indicates good prognosis, 4-6 indicates poor prognosis, and 6 indicates death.

SECONDARY OUTCOMES:
90-day mortality | 90-day
  Proportion of patients who died 90 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Guizhou Medical University Affiliated Hospital, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Q, Chen N, Ren Y, Ren S, Ye F, Zhao X, Wu G, Wang L. Morphological characteristics of CT blend sign predict hematoma expansion and outcomes in intracerebral hemorrhage in elderly patients. Front Med (Lausanne). 2024 Oct 1;11:1442724. doi: 10.3389/fmed.2024.1442724. eCollection 2024. PMID 39411190

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT05548530/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT05548530/ICF_002.pdf